CLINICAL TRIAL: NCT04470453
Title: Association Between Methotrexate Erythrocyte Polyglutamate Concentration and Biological Drug Concentration and Clinical Response in Rheumatoid Arthritis Patients Treated With Subcutaneous Injectable Methotrexate and a First Biological Drug
Acronym: POLYbio
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inclusion rate too low to meet the evaluation criterion.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19CH114; 2019-003700-12 (EudraCT Number)
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Methotrexate; Erythrocyte polyglutamate; Compliance Questionnaire Rheumatology
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with active rheumatoid arthritis (Experimental): 30 patients with active rheumatoid arthritis will be included. They will have a blood sample and Compliance Rheumatology Questionnaire (CRQ).
  Interventions: Biological: Blood sample; Diagnostic Test: CRQ
- Patients with rheumatoid arthritis into remission (Experimental): 30 patients with rheumatoid arthritis into remission will be included. They will have a blood sample and Compliance Rheumatology Questionnaire (CRQ).
  Interventions: Biological: Blood sample; Diagnostic Test: CRQ

INTERVENTIONS:
Biological: Blood sample — Blood samples will be collected for measuring PG-MTX blood concentration.
Diagnostic Test: CRQ — Compliance Rheumatology Questionnaire (CQR) is a self-administered questionnaire for to evaluate therapeutic observance during rheumatoid arthritis.
  Other Names: Compliance Rheumatology Questionnaire

SUMMARY:
The combination of methotrexate (MTX) with a biological disease-modifying antirheumatic drugs (bDMARD) is the next step in treatment with MTX monotherapy in rheumatoid arthritis (RA). Estimation of MTX and bDMARD impregnation could be performed with the erythrocyte MTX polyglutamate (MTX-PG) and bDMARD assays before to move to a second bDMARD. In RA patients treated with MTX (prescribed for at least 6 months at a stable dose for at least 3 months) in combination to a first bDMARD (prescribed since at least 3 months), an assay of MTX-PG and bDMARD will be performed in tow subsets of RA according to the level of disease activity. The first subset is active RA defined by a DAS28 (disease activity score 28)>3.2. The second one is RA in clinical remission defined by a DAS28<2.6. The main hypothesis is the association between the low concentration of MTX-PG and the clinical response of RA patients treated with subcutaneous methotrexate injection associated to a first bDMARD. Adherence to MTX will be reviewed by the Compliance Questionnaire Rheumatology (CQR) questionnaire. This assay could be useful to improve MTX management before to move to a second bDMARD.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and have social security affiliation.
* Patients followed in the Rheumatology Department at the hospital of St Etienne.
* Rheumatoid Arthritis patients in remission (Disease Activity Score 28<2.6) with methotrexate (MTX) treatment for at least 6months, and with a stable dose for 3months.
* Patients with a High Disease Activity Rheumatoid Arthritis activity (Disease Activity Score 28>3.2) with methotrexate (MTX) treatment (≥ 15 mg/week), taking MTX treatment for at least 6months with a stable subcutaneous weekly MTX injection (≥ 15 mg/week) treatment during the previous 3 months.
* Signed informed consent.

Exclusion Criteria:

* Patients treated with another conventional synthetic Disease Modifying Anti-Rheumatic Drugs (csDMARD)
* Another diagnostic than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
MTX-PG concentration | Hour 1
  To compare MTX-PG concentration in patients with active rheumatoid arthritis and patients with rheumatoid arthritis in remission

SECONDARY OUTCOMES:
metabolites dosing of MTX-PG (nmol/l) | Hour 1
  Analysis of different metabolites dosing of MTX-PG by High-performance liquid chromatography technical
Analysis of CQR score response | Hour 1
  Compliance Rheumatology Questionnaire (CRQ) is a 19-item self-administered questionnaire to measure overall patient compliance for both MTX and bDMARD treatment with 0 (bad compliance) and 100 (better compliance).

CONTACTS AND LOCATIONS:
Overall Officials: Hubert MAROTTE, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No